CLINICAL TRIAL: NCT04971798
Title: A Non-randomized, Open-label, Multi-center, Prospective Study to Evaluate the Safety and Efficacy of Intraarticular Injection of Cell-free Stem Cell-derived Extract Formulation in Patients Suffering From Knee Osteoarthritis
Brief Title: Cell-free Stem Cell-derived Extract Formulation for Knee Osteoarthritis
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: General Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GT - 2021CCM/OA
Record Dates: First submitted 2021-07-20; First posted 2021-07-21 (Actual); Last update posted 2022-07-21 (Actual); Status verified 2021-07

CONDITIONS: Osteoarthritis, Knee
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Cell-free Stem cell-derived Extract Formulation (CCM) (Experimental): Intraarticular administration of CCM
  Interventions: Biological: Cell-free Stem Cell-derived Extract Formulation (CCM)

INTERVENTIONS:
Biological: Cell-free Stem Cell-derived Extract Formulation (CCM) — Intraarticular injection

SUMMARY:
The purpose of this study is to determine the safety and efficacy of intraarticular injection of Cell-free Stem Cell-derived Extract Formulation for treatment of knee osteoarthritis symptoms.

DETAILED DESCRIPTION:
Osteoarthritis and other orthopaedic acute and degenerative conditions affect millions of people each year, resulting in significant pain and disability. Conservative modalities are limited, as they may not reverse the underlying pathology and may only provide minimal relief.

To address the limitations of traditional conservative modalities, there has been substantial interest in biologics for musculoskeletal regenerative medicine applications. The efficacy of these biologics is attributed to the presence of stem cells, growth factors (GFs), cytokines (CKs), and extracellular vesicles (EVs) including exosomes.

However, first generation biologics, specifically whole stem cell products, are not without their own inherent limitations, including establishing a reliable source with a stable phenotype, genetic instability and chromosomal aberrations, intravenous administration related toxicities caused by the physical trapping of the cells in the lung microvasculature, rejection by the host, formation of ectopic tissue, and tumorigenicity.

When considering how to harness the value of current biologics into a next generation product that can address existing limitations, it is important to consider current foundational knowledge regarding the mechanism of action of stem cell products. Recent literature regarding the beneficial effects of mesenchymal stem cells (MSCs) postulates that the mechanism of action is not due to their ability to grow and differentiate. Rather, it is secondary to their secretion of bioactive molecules such as growth factors, cytokines, and exosomes. GFs, secreted from stem cells, induce signal transduction pathways that initiate cell migration, proliferation, growth, and differentiation. CKs, similarly, can regulate inflammation, immune response, cellular differentiation, and tissue remodeling. Exosomes also are secreted by mesenchymal stem cells and act as a paracrine mediator to target cells, providing a regenerative microenvironment for damaged tissues.

As existing literature establishes that these aforementioned components of stem cells lead to regenerative responses, we have accordingly sought to establish if a sub-cellular approach to biologics can provide similar benefits while avoiding the risk profile, including immunogenicity, infection, and the potential for tumorgenicity, associated with whole stem cell products. In support of this hypothesis, recent studies have demonstrated that MSCs-derived exosomes can act as a cell-free therapeutic alternative to whole cell therapy with great regenerative potential. In addition, to the benefits by means of risk elimination, there may be further therapeutic benefits of a cellular derived therapeutic approach. For example, exosomes due to their smaller size, have the potential to migrate to target organs efficiently after, without getting trapped in the lung microvasculature. Additionally, a higher concentration of "active ingredients" can be administered directly to the patient, which may induce a larger healing response than is possible with whole stem cell therapies.

To meet these goals of improving the risk profile and therapeutic benefit of regenerative medicine, we have formulated a novel cell-free stem cell-derived extract, CCM, from human progenitor endothelial stem cells (hPESCs). Our preliminary results demonstrated presence of several GFs, anti-inflammatory CKs and EVs including exosomes in this formulation. Functionally, this formulation also significantly enhanced cell proliferation and induced stem cell migration.

The goal of this proposed study is to evaluate the safety and efficacy of intraarticular injection of this cell-free stem cell-derived extract formulation for treatment of knee osteoarthritis symptoms. We hypothesize that intraarticular administration of this cell-free stem cell-derived extract formulation is safe. We also hypothesize that patients receiving intraarticular injection of this formulation will show an improvement in their overall satisfaction, Numeric Pain rating Scale (NPRS), Patient-Reported Outcomes Measurement Information System (PROMIS) score and Knee Injury and Osteoarthritis Outcome Score (KOOS Jr.) over a period of 2-years compared to the baseline visit. Our null hypothesis is that there is no difference between baseline and follow-up visits for any outcome measures.

ELIGIBILITY:
Inclusion Criteria:

1. Be 18 years of age or older at the time of enrollment
2. Have a body mass index (BMI) of ≤ 35Kg/m2
3. Be willing and capable of giving written informed consent to participate in this clinical study based on voluntary agreement after thorough explanation of the subject's participation has been provided
4. Be willing and capable of subjective evaluation, reading and understanding written questionnaires, and reading, understanding and signing the written informed consent
5. Has been diagnosed with Mild to Moderate knee osteoarthritis (OA) in one knee only, with a Grade 2 or 3 on the Kellgren Lawrence (KL) grading scale
6. Has an average knee pain intensity ≥ 6 of the Numerical Pain Rating Scale (NPRS); Scale 0 to 10
7. Be willing to not take any knee symptom modifying drugs from baseline through the End of Study
8. Be willing and able to comply with study-related requirements, procedures, and visits
9. If female, sexually active, and of childbearing age, subject must be willing to use a reliable form of birth control throughout the duration of the study. If Male, sexually active with partners of childbearing age, must be willing to use contraceptive measures

Exclusion Criteria:

1. Has taken any pain medications, including NSAIDs, within 15 days prior to the study injection date
2. Current use of anticoagulants or history of regular use of anticoagulants
3. History of addiction to dependency producing medications or history of a substance abuse (including alcohol and illicit drugs)
4. Has mechanical knee symptoms consistent with extensive intraarticular pathology not amenable to injection therapy alone, including clinical or imaging evidence indicative of ACL, MCL, LCL, or meniscal pathology
5. Has undergone intraarticular injection of any drug including but not limited to corticosteroids or viscosupplementation in the index knee in the last 3 months
6. History of any type of surgery on the index knee
7. History of traumatic injury to the index knee within the last 3 months
8. Has planned elective knee surgery during the course of the study
9. History of organ or hematologic transplantation
10. History of rheumatoid arthritis or other autoimmune disorders
11. History of immunosuppressive medication/treatment or cancer diagnosis within the last 5 years
12. Current knee infection or history of using antibiotics for knee infection within the last 3 months
13. Has participated in another clinical study or received treatment with any investigational product within 30 days of enrollment
14. Is pregnant as determined by urine testing unless female subject is surgically sterile or post-menopausal
15. Currently breastfeeding or desires to be pregnant during the course of the study
16. Has contraindications to X-ray or MRI imaging
17. Has a diagnosis of progressive neurological disease
18. Has a diagnosis of an active psychological or psychiatric disorder
19. Has pain in other area(s) and/or medical condition(s) that could interfere with accurate pain reporting, study procedures, and/or confound evaluation of the study
20. Has unresolved major issues of secondary gain (e.g., social, financial, or legal (e.g., worker's compensation claim)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2023-01-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Treatment-emergent adverse effects as assessed by Comprehensive Metabolic Profile | 1 week
  To determine safety i.e. adverse events associated with intraarticular administration of CCM as assessed by Comprehensive metabolic profile
Treatment-emergent adverse effects as assessed by Comprehensive Metabolic Profile | 6 weeks
  To determine safety i.e. adverse events associated with intraarticular administration of CCM as assessed by Comprehensive metabolic profile
Treatment-emergent adverse effects as assessed by Comprehensive Metabolic Profile | 3 Months
  To determine safety i.e. adverse events associated with intraarticular administration of CCM as assessed by Comprehensive metabolic profile
Treatment-emergent adverse effects as assessed by Comprehensive Metabolic Profile | 6 Months
  To determine safety i.e. adverse events associated with intraarticular administration of CCM as assessed by Comprehensive metabolic profile
Treatment-emergent adverse effects as assessed by Comprehensive Metabolic Profile | 12 Months
  To determine safety i.e. adverse events associated with intraarticular administration of CCM as assessed by Comprehensive metabolic profile
Treatment-emergent adverse effects as assessed by Creatinine levels | 1 Week
  To determine safety i.e. adverse events associated with intraarticular administration of CCM as assessed by Creatinine levels
Treatment-emergent adverse effects as assessed by Creatinine levels | 6 Weeks
  To determine safety i.e. adverse events associated with intraarticular administration of CCM as assessed by Creatinine levels
Treatment-emergent adverse effects as assessed by Creatinine levels | 3 Months
  To determine safety i.e. adverse events associated with intraarticular administration of CCM as assessed by Creatinine levels
Treatment-emergent adverse effects as assessed by Creatinine levels | 6 Months
  To determine safety i.e. adverse events associated with intraarticular administration of CCM as assessed by Creatinine levels
Treatment-emergent adverse effects as assessed by Creatinine levels | 12 Months
  To determine safety i.e. adverse events associated with intraarticular administration of CCM as assessed by Creatinine levels
Treatment-emergent adverse effects as assessed by Liver Function Test | 1 Week
  To determine safety i.e. adverse events associated with intraarticular administration of CCM as assessed by Liver Function Test
Treatment-emergent adverse effects as assessed by Liver Function Test | 6 Weeks
  To determine safety i.e. adverse events associated with intraarticular administration of CCM as assessed by Liver Function Test
Treatment-emergent adverse effects as assessed by Liver Function Test | 3 Months
  To determine safety i.e. adverse events associated with intraarticular administration of CCM as assessed by Liver Function Test
Treatment-emergent adverse effects as assessed by Liver Function Test | 6 Months
  To determine safety i.e. adverse events associated with intraarticular administration of CCM as assessed by Liver Function Test
Treatment-emergent adverse effects as assessed by Liver Function Test | 12 Months
  To determine safety i.e. adverse events associated with intraarticular administration of CCM as assessed by Liver Function Test
Treatment-emergent adverse effects as assessed by Complete Blood Count | 1 Week
  To determine safety i.e. adverse events associated with intraarticular administration of CCM as assessed by Complete Blood Count
Treatment-emergent adverse effects as assessed by Complete Blood Count | 6 Weeks
  To determine safety i.e. adverse events associated with intraarticular administration of CCM as assessed by Complete Blood Count
Treatment-emergent adverse effects as assessed by Complete Blood Count | 3 Months
  To determine safety i.e. adverse events associated with intraarticular administration of CCM as assessed by Complete Blood Count
Treatment-emergent adverse effects as assessed by Complete Blood Count | 6 Months
  To determine safety i.e. adverse events associated with intraarticular administration of CCM as assessed by Complete Blood Count
Treatment-emergent adverse effects as assessed by Complete Blood Count | 12 Months
  To determine safety i.e. adverse events associated with intraarticular administration of CCM as assessed by Complete Blood Count
Treatment-emergent adverse effects as assessed by C-reactive protein | 1 Week
  To determine safety i.e. adverse events associated with intraarticular administration of CCM as assessed by C-reactive protein
Treatment-emergent adverse effects as assessed by C-reactive protein | 6 Weeks
  To determine safety i.e. adverse events associated with intraarticular administration of CCM as assessed by C-reactive protein
Treatment-emergent adverse effects as assessed by C-reactive protein | 3 Months
  To determine safety i.e. adverse events associated with intraarticular administration of CCM as assessed by C-reactive protein
Treatment-emergent adverse effects as assessed by C-reactive protein | 6 Months
  To determine safety i.e. adverse events associated with intraarticular administration of CCM as assessed by C-reactive protein
Treatment-emergent adverse effects as assessed by C-reactive protein | 12 Months
  To determine safety i.e. adverse events associated with intraarticular administration of CCM as assessed by C-reactive protein
Treatment-emergent adverse effects as assessed by Erythrocyte Sedimentation Rate | 1 Week
  To determine safety i.e. adverse events associated with intraarticular administration of CCM as assessed by Erythrocyte Sedimentation Rate
Treatment-emergent adverse effects as assessed by Erythrocyte Sedimentation Rate | 6 Weeks
  To determine safety i.e. adverse events associated with intraarticular administration of CCM as assessed by Erythrocyte Sedimentation Rate
Treatment-emergent adverse effects as assessed by Erythrocyte Sedimentation Rate | 3 Months
  To determine safety i.e. adverse events associated with intraarticular administration of CCM as assessed by Erythrocyte Sedimentation Rate
Treatment-emergent adverse effects as assessed by Erythrocyte Sedimentation Rate | 6 Months
  To determine safety i.e. adverse events associated with intraarticular administration of CCM as assessed by Erythrocyte Sedimentation Rate
Treatment-emergent adverse effects as assessed by Erythrocyte Sedimentation Rate | 12 Months
  To determine safety i.e. adverse events associated with intraarticular administration of CCM as assessed by Erythrocyte Sedimentation Rate
Treatment-emergent adverse effects as assessed by T, B and NK Cell Lymphocyte subsets | 1 Week
  To determine safety i.e. adverse events associated with intraarticular administration of CCM as assessed by T, B and NK Cell Lymphocyte subsets
Treatment-emergent adverse effects as assessed by T, B and NK Cell Lymphocyte subsets | 6 Weeks
  To determine safety i.e. adverse events associated with intraarticular administration of CCM as assessed by T, B and NK Cell Lymphocyte subsets
Treatment-emergent adverse effects as assessed by T, B and NK Cell Lymphocyte subsets | 3 Months
  To determine safety i.e. adverse events associated with intraarticular administration of CCM as assessed by T, B and NK Cell Lymphocyte subsets
Treatment-emergent adverse effects as assessed by T, B and NK Cell Lymphocyte subsets | 6 Months
  To determine safety i.e. adverse events associated with intraarticular administration of CCM as assessed by T, B and NK Cell Lymphocyte subsets
Treatment-emergent adverse effects as assessed by T, B and NK Cell Lymphocyte subsets | 12 Months
  To determine safety i.e. adverse events associated with intraarticular administration of CCM as assessed by T, B and NK Cell Lymphocyte subsets
Treatment-emergent adverse effects as assessed by Serum IgG, IgA, IgM and IgE levels | 1 Week
  To determine safety i.e. adverse events associated with intraarticular administration of CCM as assessed by Serum IgG, IgA, IgM and IgE levels
Treatment-emergent adverse effects as assessed by Serum IgG, IgA, IgM and IgE levels | 6 Weeks
  To determine safety i.e. adverse events associated with intraarticular administration of CCM as assessed by Serum IgG, IgA, IgM and IgE levels
Treatment-emergent adverse effects as assessed by Serum IgG, IgA, IgM and IgE levels | 3 Months
  To determine safety i.e. adverse events associated with intraarticular administration of CCM as assessed by Serum IgG, IgA, IgM and IgE levels
Treatment-emergent adverse effects as assessed by Serum IgG, IgA, IgM and IgE levels | 6 Months
  To determine safety i.e. adverse events associated with intraarticular administration of CCM as assessed by Serum IgG, IgA, IgM and IgE levels
Treatment-emergent adverse effects as assessed by Serum IgG, IgA, IgM and IgE levels | 12 Months
  To determine safety i.e. adverse events associated with intraarticular administration of CCM as assessed by Serum IgG, IgA, IgM and IgE levels

SECONDARY OUTCOMES:
Change in patient reported outcome measures, Numeric Pain Rating Scale | Change from baseline to immediately after injection
  To determine change in patient reported outcome measure, Numeric Pain Rating Scale (NPRS). A decrease in score indicates improvement.
Change in patient reported outcome measures, Numeric Pain Rating Scale | Change from baseline to 24 hours after injection
  To determine change in patient reported outcome measure, Numeric Pain Rating Scale (NPRS). A decrease in score indicates improvement.
Change in patient reported outcome measures, Numeric Pain Rating Scale | Change from baseline to 48 hours after injection
  To determine change in patient reported outcome measure, Numeric Pain Rating Scale (NPRS). A decrease in score indicates improvement.
Change in patient reported outcome measures, Numeric Pain Rating Scale | Change from baseline to 1 week after injection
  To determine change in patient reported outcome measure, Numeric Pain Rating Scale (NPRS). A decrease in score indicates improvement.
Change in patient reported outcome measures, Numeric Pain Rating Scale | Change from baseline to 6 weeks after injection
  To determine change in patient reported outcome measure, Numeric Pain Rating Scale (NPRS). A decrease in score indicates improvement.
Change in patient reported outcome measures, Numeric Pain Rating Scale | Change from baseline to 3 months after injection
  To determine change in patient reported outcome measure, Numeric Pain Rating Scale (NPRS). A decrease in score indicates improvement.
Change in patient reported outcome measures, Numeric Pain Rating Scale | Change from baseline to 6 months after injection
  To determine change in patient reported outcome measure, Numeric Pain Rating Scale (NPRS). A decrease in score indicates improvement.
Change in patient reported outcome measures, Numeric Pain Rating Scale | Change from baseline to 12 months after injection
  To determine change in patient reported outcome measure, Numeric Pain Rating Scale (NPRS). A decrease in score indicates improvement.
Change in patient reported outcome measures, Numeric Pain Rating Scale | Change from baseline to 18 months after injection
  To determine change in patient reported outcome measure, Numeric Pain Rating Scale (NPRS). A decrease in score indicates improvement.
Change in patient reported outcome measures, Numeric Pain Rating Scale | Change from baseline to 24 months after injection
  To determine change in patient reported outcome measure, Numeric Pain Rating Scale (NPRS). A decrease in score indicates improvement.
Change in patient reported outcome measures, Knee Injury and Osteoarthritis Outcome Score Jr. | Change from baseline to 1 week after injection
  To determine change in patient reported outcome measure, Knee Injury and Osteoarthritis Outcome Score Jr. (KOOS Jr.). An increase in score indicates improvement.
Change in patient reported outcome measures, Knee Injury and Osteoarthritis Outcome Score Jr. | Change from baseline to 6 weeks after injection
  To determine change in patient reported outcome measure, Knee Injury and Osteoarthritis Outcome Score Jr. (KOOS Jr.). An increase in score indicates improvement.
Change in patient reported outcome measures, Knee Injury and Osteoarthritis Outcome Score Jr. | Change from baseline to 3 months after injection
  To determine change in patient reported outcome measure, Knee Injury and Osteoarthritis Outcome Score Jr. (KOOS Jr.). An increase in score indicates improvement.
Change in patient reported outcome measures, Knee Injury and Osteoarthritis Outcome Score Jr. | Change from baseline to 6 months after injection
  To determine change in patient reported outcome measure, Knee Injury and Osteoarthritis Outcome Score Jr. (KOOS Jr.). An increase in score indicates improvement.
Change in patient reported outcome measures, Knee Injury and Osteoarthritis Outcome Score Jr. | Change from baseline to 12 months after injection
  To determine change in patient reported outcome measure, Knee Injury and Osteoarthritis Outcome Score Jr. (KOOS Jr.). An increase in score indicates improvement.
Change in patient reported outcome measures, Knee Injury and Osteoarthritis Outcome Score Jr. | Change from baseline to 18 months after injection
  To determine change in patient reported outcome measure, Knee Injury and Osteoarthritis Outcome Score Jr. (KOOS Jr.). An increase in score indicates improvement.
Change in patient reported outcome measures, Knee Injury and Osteoarthritis Outcome Score Jr. | Change from baseline to 24 months after injection
  To determine change in patient reported outcome measure, Knee Injury and Osteoarthritis Outcome Score Jr. (KOOS Jr.). An increase in score indicates improvement.
Change in patient reported outcome measures, Patient-Reported Outcomes Measurement Information System (PROMIS) score. | Change from baseline to 1 week after injection
  To determine change in patient reported outcome measure, Patient-Reported Outcomes Measurement Information System (PROMIS) score. An increase in score indicates improvement.
Change in patient reported outcome measures, Patient-Reported Outcomes Measurement Information System (PROMIS) score. | Change from baseline to 6 weeks after injection
  To determine change in patient reported outcome measure, Patient-Reported Outcomes Measurement Information System (PROMIS) score. An increase in score indicates improvement.
Change in patient reported outcome measures, Patient-Reported Outcomes Measurement Information System (PROMIS) score. | Change from baseline to 3 months after injection
  To determine change in patient reported outcome measure, Patient-Reported Outcomes Measurement Information System (PROMIS) score. An increase in score indicates improvement.
Change in patient reported outcome measures, Patient-Reported Outcomes Measurement Information System (PROMIS) score. | Change from baseline to 6 months after injection
  To determine change in patient reported outcome measure, Patient-Reported Outcomes Measurement Information System (PROMIS) score. An increase in score indicates improvement.
Change in patient reported outcome measures, Patient-Reported Outcomes Measurement Information System (PROMIS) score. | Change from baseline to 12 months after injection
  To determine change in patient reported outcome measure, Patient-Reported Outcomes Measurement Information System (PROMIS) score. An increase in score indicates improvement.
Change in patient reported outcome measures, Patient-Reported Outcomes Measurement Information System (PROMIS) score. | Change from baseline to 18 months after injection
  To determine change in patient reported outcome measure, Patient-Reported Outcomes Measurement Information System (PROMIS) score. An increase in score indicates improvement.
Change in patient reported outcome measures, Patient-Reported Outcomes Measurement Information System (PROMIS) score. | Change from baseline to 24 months after injection
  To determine change in patient reported outcome measure, Patient-Reported Outcomes Measurement Information System (PROMIS) score. An increase in score indicates improvement.
Patient Satisfaction via 5-point Likert Scale | 1 Week after injection
  To determine patient satisfaction via 5-point Likert Scale. An increase in score indicates improvement.
Patient Satisfaction via 5-point Likert Scale | 6 Weeks after injection
  To determine patient satisfaction via 5-point Likert Scale. An increase in score indicates improvement.
Patient Satisfaction via 5-point Likert Scale | 3 Months after injection
  To determine patient satisfaction via 5-point Likert Scale. An increase in score indicates improvement.
Patient Satisfaction via 5-point Likert Scale | 6 Months after injection
  To determine patient satisfaction via 5-point Likert Scale. An increase in score indicates improvement.
Patient Satisfaction via 5-point Likert Scale | 12 Months after injection
  To determine patient satisfaction via 5-point Likert Scale. An increase in score indicates improvement.
Patient Satisfaction via 5-point Likert Scale | 18 Months after injection
  To determine patient satisfaction via 5-point Likert Scale. An increase in score indicates improvement.
Patient Satisfaction via 5-point Likert Scale | 24 Months after injection
  To determine patient satisfaction via 5-point Likert Scale. An increase in score indicates improvement.
Patient Satisfaction via Single Assessment Numeric Evaluation (SANE) | Change from baseline to 1 week after injection
  To determine patient satisfaction via Single Assessment Numeric Evaluation (SANE). An increase in score indicates improvement.
Patient Satisfaction via Single Assessment Numeric Evaluation (SANE) | Change from baseline to 6 weeks after injection
  To determine patient satisfaction via Single Assessment Numeric Evaluation (SANE). An increase in score indicates improvement.
Patient Satisfaction via Single Assessment Numeric Evaluation (SANE) | Change from baseline to 3 months after injection
  To determine patient satisfaction via Single Assessment Numeric Evaluation (SANE). An increase in score indicates improvement.
Patient Satisfaction via Single Assessment Numeric Evaluation (SANE) | Change from baseline to 6 months after injection
  To determine patient satisfaction via Single Assessment Numeric Evaluation (SANE). An increase in score indicates improvement.
Patient Satisfaction via Single Assessment Numeric Evaluation (SANE) | Change from baseline to 12 months after injection
  To determine patient satisfaction via Single Assessment Numeric Evaluation (SANE). An increase in score indicates improvement.
Patient Satisfaction via Single Assessment Numeric Evaluation (SANE) | Change from baseline to 18 months after injection
  To determine patient satisfaction via Single Assessment Numeric Evaluation (SANE). An increase in score indicates improvement.
Patient Satisfaction via Single Assessment Numeric Evaluation (SANE) | Change from baseline to 24 months after injection
  To determine patient satisfaction via Single Assessment Numeric Evaluation (SANE). An increase in score indicates improvement.
Patient Satisfaction via 36-item short form survey (SF36) | Change from baseline to 3 months after injection
  To determine patient satisfaction via 36-item short form survey (SF36). An increase in score indicates improvement.
Patient Satisfaction via 36-item short form survey (SF36) | Change from baseline to 6 months after injection
  To determine patient satisfaction via 36-item short form survey (SF36). An increase in score indicates improvement.
Patient Satisfaction via 36-item short form survey (SF36) | Change from baseline to 12 months after injection
  To determine patient satisfaction via 36-item short form survey (SF36). An increase in score indicates improvement.
Patient Satisfaction via 36-item short form survey (SF36) | Change from baseline to 18 months after injection
  To determine patient satisfaction via 36-item short form survey (SF36). An increase in score indicates improvement.
Patient Satisfaction via 36-item short form survey (SF36) | Change from baseline to 24 months after injection
  To determine patient satisfaction via 36-item short form survey (SF36). An increase in score indicates improvement.
Cartilage Formation | Change from baseline to 12 months after injection
  To assess cartilage formation via MOCART (Magnetic Resonance Observation of Cartilage Repair Tissue). An increase in score indicates improvement.
Cartilage Formation | Change from baseline to 24 months after injection
  To assess cartilage formation via MOCART (Magnetic Resonance Observation of Cartilage Repair Tissue). An increase in score indicates improvement.

CONTACTS AND LOCATIONS:
Overall Officials: Craig Cady, PhD, Study Director — General Therapeutics

REFERENCES:
- [Derived] Gupta A, Maffulli N, Rodriguez HC, Mistovich RJ, Delfino K, Cady C, Fauser AM, Cundiff ED, Martinez MA, Potty AG. Cell-free stem cell-derived extract formulation for treatment of knee osteoarthritis: study protocol for a preliminary non-randomized, open-label, multi-center feasibility and safety study. J Orthop Surg Res. 2021 Aug 20;16(1):514. doi: 10.1186/s13018-021-02672-3. PMID 34416898